CLINICAL TRIAL: NCT00002463
Title: Phase II Study of Methotrexate, Mechlorethamine, Vincristine, Prednisone, and Procarbazine (MMOPP) as Primary Therapy in Infants or Young Children With Primitive Neuroectodermal Tumors or High-Grade Astrocytoma
Brief Title: Combination Chemotherapy in Treating Children With Astrocytomas and Primitive Neuroectodermal Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P88-006; P30CA016672 (NIH); MDA-P-88006; NCI-V89-0125; CDR0000075917 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 1999-11-01; First posted 2004-04-22 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: childhood infratentorial ependymoma; childhood low-grade cerebral astrocytoma; childhood low-grade cerebellar astrocytoma; childhood supratentorial ependymoma; childhood high-grade cerebral astrocytoma; untreated childhood supratentorial primitive neuroectodermal tumor; untreated childhood cerebellar astrocytoma; untreated childhood medulloblastoma; untreated childhood visual pathway and hypothalamic glioma; newly diagnosed childhood ependymoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma | interventions — MOPP protocol; Leucovorin; Mechlorethamine; Methotrexate; Prednisone; Procarbazine; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Combination Chemotherapy (Experimental): Methotrexate, Mechlorethamine, Vincristine, Prednisone, and Procarbazine
  Interventions: Drug: MOPP Regimen; Drug: Leucovorin Calcium; Drug: Mechlorethamine Hydrochloride; Drug: Methotrexate; Drug: Prednisone; Drug: Procarbazine Hydrochloride; Drug: Vincristine Sulfate; Procedure: Conventional Surgery

INTERVENTIONS:
Drug: MOPP Regimen — Methotrexate, Mechlorethamine, Vincristine, Prednisone, and Procarbazine (MMOPP)
Drug: Leucovorin Calcium
Drug: Mechlorethamine Hydrochloride
Drug: Methotrexate
Drug: Prednisone
Drug: Procarbazine Hydrochloride
Drug: Vincristine Sulfate
Procedure: Conventional Surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of methotrexate, mechlorethamine, vincristine, procarbazine, and prednisone in treating children with astrocytomas or primitive neuroectodermal tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of high-dose methotrexate (HMTX) in combination with mechlorethamine, vincristine, prednisone, and procarbazine (MOPP) in infants or young children with primitive neuroectodermal tumors (PNET) (including medulloblastoma, anaplastic ependymoma, ependymoblastoma, or pineoblastoma) or high-grade astrocytoma. II. Determine whether the addition of HMTX to MOPP (MMOPP) improves the continuous complete response rate of MOPP alone and eliminates the need for salvage with radiotherapy in these patients. III. Determine the ability of MMOPP to provide neuroaxis prophylaxis or to treat spinal metastasis without radiotherapy in infants or young children with PNET. IV. Determine the toxicity of this regimen in terms of neurologic and neuropsychologic sequelae, growth, and development in these patients. V. Correlate the efficacy of this regimen with the histopathologic diagnosis of these patients. VI. Determine the optimum method for radiographic evaluation of spinal cord disease in patients with PNET. VII. Determine the utility of sequential spinal cord radiography as a means of monitoring PNET in these patients.

OUTLINE: Patients undergo maximum tumor debulking. Patients who have undergone incomplete resection proceed to induction. Patients with a primary diagnosis of primitive neuroectodermal and pineal tumors or glioblastoma multiforme who have undergone total resection proceed to induction. Induction: Patients receive high dose methotrexate (HMTX) IV over 6 hours on day 1. Beginning 3 hours after completion of HMTX infusion, leucovorin calcium (CF) is administered IV over 30 minutes every 3 hours for 9 doses. Beginning 3 hours after completion of the last CF infusion, oral CF is administered every 6 hours for 8 doses. Patients receive a second HMTX infusion beginning 1 week after completion of the first HMTX infusion. Beginning 1 week after completion of the second HMTX infusion, patients receive mechlorethamine IV and vincristine IV on days 1 and 8, oral procarbazine and oral prednisone on days 1-10, and tapered doses of prednisone on days 11-13 (MOPP). Maintenance: Beginning 4 weeks after initiating the first course of MOPP, patients receive HMTX on day 1 and MOPP beginning on day 4. Treatment continues every 31 days in the absence of disease progression or unacceptable toxicity. After 1 year or 14 doses of HMTX, whichever occurs first, HMTX is discontinued and treatment with MOPP alone continues every 4 weeks in the absence of disease progression or unacceptable toxicity. Treatment is discontinued after 2 years if the patient is in continuous complete remission.

PROJECTED ACCRUAL: A total of 5-25 patients will be accrued for this study within 24-30 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven previously untreated (except surgically) primitive neuroectodermal tumors (including medulloblastoma, anaplastic ependymoma, ependymoblastoma, or pineoblastoma) or high-grade astrocytomas Low-grade astrocytomas or optic tract tumors that are incompletely resected and have a progressive course not amenable to further surgery may also be allowed Evaluable disease by MRI, CT scan, or CT myelography

PATIENT CHARACTERISTICS: Age: Under 4 years Performance status: Not specified Life expectancy: At least 12 weeks Hematopoietic: Absolute granulocyte count greater than 1,500/mm3 WBC greater than 4,000/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin less than 1.5 mg/dL SGPT less than 90 IU/dL Renal: Creatinine clearance greater than 80 mL/min

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent immunotherapy Chemotherapy: No prior mechlorethamine, vincristine, procarbazine, and prednisone (MOPP) No prior high-dose methotrexate No other concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: No concurrent radiotherapy Surgery: See Disease Characteristics Other: Recovered from acute toxic effects of any prior therapy Must be on a tyramine-free diet during procarbazine administration

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 1989-02; Primary Completion 2007-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Number of Patient with Overall Response | Every 31 days

CONTACTS AND LOCATIONS:
Overall Officials: Joann Ater, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas - MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Result] Ater J, Worth L, Bruner J, et al.: Young children treated with MOPP or methotrexate-MOP for medulloblastoma: identification of a subset of patients with good prognosis. [Abstract] Proceedings of the American Society of Clinical Oncology 14: A-1397, 1995.
- [Result] Ater JL, van Eys J, Yung WK, et al.: Response to methotrexate, mechlorethamine, vincristine, procarbazine, and prednizone (MMOPP) for brain tumors. [Abstract] Proceedings of the American Society of Clinical Oncology 10: A-370, 125, 1991.